CLINICAL TRIAL: NCT00397007
Title: Evaluation of Psychological and Psychophysiological Effects of a Biofeedback-based Cognitive-behavioral Psychotherapy for Chronic Tinnitus-sufferers
Brief Title: Psychophysiological Treatment of Chronic Tinnitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Winfried Rief, Professor Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RI 574/12-1
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Tinnitus
Keywords: tinnitus; biofeedback; psychophysiological reactivity; intervention
MeSH Terms: conditions — Tinnitus

INTERVENTIONS:
Behavioral: Biofeedback-based cognitive-behavioural intervention

SUMMARY:
The study aims to develop and to evaluate a psychophysiological intervention for distressing chronic tinnitus. Therefore 100 people suffering from chronic tinnitus are randomly assigned to either an intervention-group, receiving 12 sessions of a psychophysiological oriented intervention, or to a waiting-list-group, who are waiting for a comparable time period. Afterwards, patients of the waiting-list-group also receive intervention. The effects of the intervention on severity, distress and perceived loudness of the tinnitus as well as on other psychological variables like depression or self-efficacy are evaluated through comparing the results of the intervention group with those of the waiting-list-group.

Additionally the psychophysiological reactivity under different stress-conditions is measured before and after intervention or waiting. Therefore the activity of the muscles of head and shoulders (EMG) as well as the skin temperature and skin conductance are measured. It is hypothesized that patients with stronger psychophysiological reactivity benefit more from an psychophysiological intervention.

DETAILED DESCRIPTION:
The study aims to develop and to evaluate a psychophysiological intervention for distressing chronic tinnitus. Therefore 100 people suffering from chronic tinnitus are randomly assigned to either an intervention-group, receiving 12 sessions of a psychophysiological oriented intervention, or to a waiting-list-group, who are waiting for a comparable time period. Afterwards, patients of the waiting-list-group also receive intervention. The effects of the intervention on severity, distress and perceived loudness of the tinnitus as well as on other psychological variables like depression or self-efficacy are evaluated through comparing the results of the intervention group with those of the waiting-list-group.

Additionally the psychophysiological reactivity under different stress-conditions is measured before and after intervention or waiting. Therefore the activity of the muscles of head and shoulders (EMG) as well as the skin temperature and skin conductance are measured. It is hypothesized that patients with stronger psychophysiological reactivity benefit more from an psychophysiological intervention.

Further aims of the study are 1) to compare the muscle activity of the tinnitus-patients with those from healthy controls, because till now no study investigated if tinnitus-patients effectively present higher muscle activity in head and shoulders than healthy people and 2) to evaluate the influence of the subjective illness perceptions on the intervention-outcome, because it is hypothesized that patients with more somatic illness perceptions benefit more from a psychophysiological intervention than patients with rather psychological illness perceptions.

ELIGIBILITY:
Inclusion Criteria:

* 100 subjects with distressing and chronic tinnitus (for at least 6 month)
* age: 16-75 years
* sufficient language skills

plus

* 50 healthy control-subjects
* without tinnitus or other hearing disease

Exclusion Criteria (for both):

* tinnitus as a result of medical disease (e.g.Meniere's disease)
* attendance in the previous study
* psychosis or dementia

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2005-05; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Tinnitus Questionnaire German Version
Tinnitus diary

SECONDARY OUTCOMES:
Symptom Check List
Beck Depression Inventory
Illness perception questionnaire
Pain disability index
Generalized self efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Study Director — Philipps University Marburg
Locations (1):
- Philipps-University Marburg, Faculty of Psychology, Marburg, Germany

REFERENCES:
- [Background] Rief W, Weise C, Kley N, Martin A. Psychophysiologic treatment of chronic tinnitus: a randomized clinical trial. Psychosom Med. 2005 Sep-Oct;67(5):833-8. doi: 10.1097/01.psy.0000174174.38908.c6. PMID 16204446
- [Result] Heinecke K, Weise C, Schwarz K, Rief W. Physiological and psychological stress reactivity in chronic tinnitus. J Behav Med. 2008 Jun;31(3):179-88. doi: 10.1007/s10865-007-9145-0. Epub 2008 Jan 12. PMID 18193350
- [Result] Weise, C, Heinecke, K, & Rief, W . Biofeedback bei chronischem Tinnitus - Behandlungsleitfaden und vorläufige Ergebnisse zu Wirksamkeit und Akzeptanz [Biofeedback for chronic tinnitus - Treatment guidelines and preliminary results regarding their efficacy and acceptance]. Verhaltenstherapie 17(4): 220-230, 2007.
- [Derived] Weise C, Heinecke K, Rief W. Biofeedback-based behavioral treatment for chronic tinnitus: results of a randomized controlled trial. J Consult Clin Psychol. 2008 Dec;76(6):1046-57. doi: 10.1037/a0013811. PMID 19045972
- [Derived] Weise C, Heinecke K, Rief W. Stability of physiological variables in chronic tinnitus sufferers. Appl Psychophysiol Biofeedback. 2008 Sep;33(3):149-59. doi: 10.1007/s10484-008-9058-x. Epub 2008 Jul 4. PMID 18600443